CLINICAL TRIAL: NCT01963832
Title: RCT of a Neuroplasticity Agent and CI Therapy for Severe Arm Paresis After Stroke
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: not funded
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F130410007
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2014-12

CONDITIONS: Severe Stroke With Affected Arm Motor Function
Keywords: stroke; Fluoxetine (FLX); eCIMT; Central Nervous System
MeSH Terms: conditions — Stroke | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- eCMIT and Fluoxetine (Experimental): expanded form of Constraint Induced Movement Therapy (eCIMT) combined with Fluoxetine (FLX)
  Interventions: Drug: Fluoxetine; Procedure: eCMIT
- eCIMT and placebo (Experimental): expanded form of Constraint Induced Movement Therapy (eCIMT) combined with placebo
  Interventions: Drug: Fluoxetine; Drug: Placebo
- Usual care and fluoxetine (Experimental): Ususal physical care combined with Fluoxetine (FLX)
  Interventions: Drug: Fluoxetine; Procedure: Usual Care
- Usual care and placebo (Experimental): Usual physical care combined with placebo
  Interventions: Drug: Placebo; Procedure: Usual Care

INTERVENTIONS:
Drug: Fluoxetine
  Arms: Usual care and fluoxetine; eCIMT and placebo; eCMIT and Fluoxetine
Drug: Placebo
  Arms: Usual care and placebo; eCIMT and placebo
Procedure: eCMIT
  Arms: eCMIT and Fluoxetine
Procedure: Usual Care
  Arms: Usual care and fluoxetine; Usual care and placebo

SUMMARY:
Stroke patients who have little or no voluntary movement in the hand on the more affected side of their body more than one year after stroke have few treatment options. This project proposes to test the efficacy of a form of Constraint-Induced Movement therapy designed for patients with such severe impairment in conjunction with an agent, fluoxetine, which has been shown in some studies to enhance brain neuroplasticity in response to training. Constraint-Induced Movement therapy, which is abbreviated CIMT, is a form of physical rehabilitation based on basic research in neuroscience and behavioral science. If the project is successful, an efficacious, evidence-based therapy will become available to stroke patients for what is now a largely untreated condition

ELIGIBILITY:
Inclusion Criteria:

* Motor criteria determinations will be made with the subject sitting. The more-affected forearm will be resting on a supporting surface (e.g., arm of a chair) to allow for maximum wrist flexion with gravity.
* The minimum motor criterion (MMC) for inclusion in Grade 5 (severe impairment) will be ability to:

  * initiate extension against gravity at the wrist or at least one digit,
  * initiate extension and flexion at the elbow,
  * actively move the shoulder ≥ 30° in flexion, abduction, or scaption
* The MMC for inclusion in Grade 4 (moderately severe impairment) will be ability to actively:

  * extend at least two fingers more than 0° but less than < 10°,
  * extend or abduct thumb ≥ 10°
  * extend wrist ≥ 10° from a fully flexed starting position,
  * extend elbow ≥ 20° from a 90° flexed starting position,
  * flex and abduct shoulder > 45°.
* Stroke patients who can extend at least two fingers ≥ 10° at the metacarpophalangeal (MCP) joint and either the proximal or distal interphalangeal (PIP or DIP) joint will be excluded.
* Additional inclusion criteria are:

  * must score ≤ 4 on the Modified Ashworth Scale (23)116 for all more-affected arm joints
  * meet the following passive range of movement criteria:

    * ≥ 90° shoulder flexion,
    * ≥ 90° shoulder abduction,
    * ≥ 45° shoulder external rotation,
    * ≤ 30° short of normal elbow extension, forearm supination to at least neutral,
    * forearm pronation 45° or more from neutral,
    * ≤ 35° short of normal wrist extension,
    * ≤ 35° short of normal MCP extension on all the digits.

Exclusion Criteria:

* Less than 1 year post-stroke.
* Frailty or insufficient stamina to carry out the requirements of the therapy (based on clinical judgment).
* Ferrous metal in body or medical complications or psychological problems that would prohibit receiving an MRI.
* Positive pregnancy test for women of child-bearing age since 3T MRI is contraindicated for pregnant women.
* Other neurological or musculoskeletal conditions affecting UE function.
* Medication will not be exclusionary except in the following cases: a. participation in any experimental drug study, b. Botox injections to the more-affected UE < 3 months prior to enrollment, c. Baclofen or Dantrium taken orally at the time of study, d. fluoxetine or other antidepressant with SSRI-like properties taken < 3 months prior to enrollment, e. any agents that would contraindicate concurrent fluoxetine. If subjects are on other medications, the medications will be recorded and the possible effect on treatment outcome will be analyzed separately.
* Moderate or greater depressive symptoms as indicated by a score > 30/63 on the Beck Depression Inventory (24,25).117, 118
* Concurrent participation in any formal physical rehabilitation program or clinical trial.
* Excessive pain in any joint of the more-affected arm that could limit ability to cooperate with the intervention (based on clinical judgment).
* Serious cognitive deficits manifested by a Folstein Mini-Mental State Examination (MMSE) score ≤ 24 (26).119
* Inadequate ability to follow test instructions as indicated by a Token Test of the Multilingual Aphasia Examination score ≤ 36 (27).120
* Serious, uncontrolled medical problems as judged by the Medical Director (e.g., severe rheumatoid arthritis, serious joint deformity of arthritic origin, symptomatic cancer or renal disease, any end-stage pulmonary or cardiovascular disease, senility or a deteriorated condition due to age, uncontrolled epilepsy).
* Motor problems that are not primarily unilateral.
* Poor motivation to participate in the study (if a person is only marginally interested, he/she is a bad risk as a subject).
* Less than 40 years old.
* Previous CIMT.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2020-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Grade 4/5 Motor Activity Log (MAL) Arm Use Scale | baseline to 90 days
  This is a structured interview. Patients and family caregivers, if available, are asked to rate how well and how much the stroke survivor has used his or her more-affected arm on 30 upper-extremity tasks outside of the treatment setting over a specified period. The test score is the mean of the item scores. The primary outcome will be change on this instrument from pre- to post-treatment.

SECONDARY OUTCOMES:
Grade 4/5 MAL Arm Use scale | baseline to 12 months after therapy
  See primary outcome.
Grade 4/5 Wolf Motor Function Test Performance Rate score | baseline to 90 days
  This is a laboratory motor performance test. Patients are asked to complete the items are rapidly as possible. Performance is timed and converted to a rate (repetitions/60 s). The test score is the mean of the item scores.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States